CLINICAL TRIAL: NCT03121404
Title: Mechanisms of Malnutrition in Cirrhosis With Portosystemic Shunting
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff Physician, The Cleveland Clinic
Other Study IDs: 08-546
Record Dates: First submitted 2017-04-12; First posted 2017-04-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cirrhosis Patient: Patients will be identified from the transplant list. Inclusion criteria will be all subjects with cirrhosis of any etiology who will undergo liver transplantation. . Rectus abdominis muscle biopsy will be obtained directly after induction of anesthesia for the procedure. In addition patients will have anthropometric measurements taken within 2 weeks of surgery. For the cirrhotic patients this includes hand grip test and dual energy x-ray absorption (DEXA).
  Interventions: Procedure: Rectus abdominis muscle biopsy
- Healthy Controls: Controls will be identified from the abdominal surgery operating room lists at Cleveland Clinic. Rectus abdominis muscle biopsy will be obtained directly after induction of anesthesia for the procedure. In addition patients will have anthropometric measurements taken within 2 weeks of surgery which will not include DEXA or hand grip test.
  Interventions: Procedure: Rectus abdominis muscle biopsy

INTERVENTIONS:
Procedure: Rectus abdominis muscle biopsy — Patients who will already be having either liver transplant surgery or abdominal surgery will have a biopsy of their rectus abdominis muscle during the time of surgery.

SUMMARY:
Cirrhosis is characterized by loss of muscle as well as fat mass, which increases morbidity and mortality before, during, and after liver transplantation. A common mechanism for the reduced muscle and fat mass in cirrhosis is an increased expression of the TGF (transforming growth factor)beta superfamily member, myostatin, in the muscle and adipose tissue. The present study will examine the expression of myostatin, its receptor and intracellular signaling pathways in the skeletal muscle and mesenteric adipose tissue in cirrhotic patients undergoing liver transplantation as compared to healthy controls undergoing planned abdominal surgery. 16 cirrhotic patients will be identified from the transplant list, and 16 healthy controls from outpatient surgery lists. Nutritional assessment will be performed, including anthropometry (triceps skinfold thickness, mid arm circumference), dual energy x-ray absorptiometry (DEXA), and bioelectrical impedance analysis (BIA). Rectus abdominis muscle tissue and omental fat tissue will be harvested in the operating room, and the expression of signaling proteins involved in skeletal muscle protein synthesis will be quantified. The investigator will also quantify the expression of genes involved in lipolysis and lipid synthesis. The investigator anticipates that the expression of myostatin will be higher in the skeletal muscle and adipose tissue of cirrhotics as compared to controls. There will be a reduction in the expression of the signaling proteins that regulate skeletal muscle protein synthesis, as well as the expression of genes regulating lipogenesis. The increased expression of myostatin will also correlate with reduced anthropometric and DEXA measurements of lean body mass and fat mass.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Patients undergoing abdominal surgery (liver transplantation or other surgery)

Control

1. non liver transplant donor
2. Elective abdominal surgery (cholecystectomy, diverticulosis, acute gastrointestinal bleeding in the absence of exclusion criteria)

Exclusion Criteria:

* Exclusion criteria (all subjects)
* Average daily alcohol intake > 20 g in women and > 30 g in men
* Diabetes or a fasting serum glucose > 100 mg/dL
* Hyper- / hypo- thyroidism
* Renal disease with serum creatinine > 1.4 mg/dL
* Folate or vitamin B12 deficiency
* Active intravenous drug use
* History of bowel surgery or gastric bypass surgery
* Medications/supplements that affect fat mass or protein mass (creatine, glucocorticoids)
* Pregnancy
* Chronic diseases that result in cachexia (renal, cardiac, pulmonary, hematologic, cancer)
* Hepatocellular cancer

Exclusion criteria (controls)

* Evidence of malnutrition as quantified by triceps skinfold thickness, mid arm muscle area and creatinine height index)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from the Cleveland Clinic transplant list. All subjects with cirrhosis of any etiology who will undergo liver transplantation will make up the group of cirrhosis patients. The controls will be patients without cirrhosis that are undergoing abdominal surgery will be identified from the operating room list at Cleveland Clinic. Rectus abdominis muscle biopsies will be obtained directly after induction of anesthesia for the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-11-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the difference in myostatin expression between healthy control and cirrhosis patients | 15 minute biopsy
  The primary outcome of this study is to determine the difference in expression of myostatin in skeletal muscle in a one time biopsy of the Rectus abdominis muscle between healthy controls and cirrhotic patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States